CLINICAL TRIAL: NCT04696302
Title: Focus of Attention Effects on Motor Performance and Learning in Individuals Post Stroke During Seated Lateral Weight Shifting: A Two-phase Feasibility Study
Brief Title: Focus of Attention in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Carolina University (Other)
Collaborators: Mission Health System, Asheville, NC (Other)
Responsible Party: Principal Investigator, Ashley Hyatt, Assistant Professor of Physical Therapy, Western Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 949671-4
Record Dates: First submitted 2020-12-16; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Cerebrovascular Accident
Keywords: Focus of attention; Motor learning; Seated weight shifting
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two independent groups measured at 4 timepoints, baseline, acquisition, short-term, and long-term retention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded from whether they were in control or experimental group and statistician was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focus of attention in individuals post chronic stroke during seated lateral weight shifting (Experimental): Feasibility study
  Interventions: Behavioral: Focus of attention
- Focus of attention in individuals post acute stroke during seated lateral weight shifting (Experimental): Feasibility study
  Interventions: Behavioral: Focus of attention

INTERVENTIONS:
Behavioral: Focus of attention — Individuals were asked to laterally weight shift while seated with either internal focus or external focus instructions.
  Other Names: Seated lateral weight shifting

SUMMARY:
This two phase feasibility study looked at the feasibility of conducting a clinical trial in the outpatient and inpatient rehab setting exploring how individuals post stroke respond to different focus of attention cues. Focus of attention refers to whether individuals in are thinking about how their body is moving, internal focus, or on the effect their body has on the environment, external focus, during motor task. This trial will specifically look at the effect focus of attention has on motor performance and learning in individuals post stroke during lateral seated weight shifting task.

DETAILED DESCRIPTION:
This was a two phase feasibility study exploring appropriate management, setting, participants including inclusion and exclusion criteria, attrition rates, protocol, and retention. Outcome data for each stage were collected during baseline, acquisition, short-term, and long-term retention.

There were two primary objectives of this two phase feasibility study. The first was to uncover some potential short comings in research designs used in this area. The second was to explore the feasibility of a study in both the chronic and acute stroke populations in a rural community. Topics of feasibility include recruitment, retention, and specific inclusion and exclusion criteria. Extending the work by Muckel and Merholz, this feasibility study examined performance of individuals post stroke during a seated lateral weight shifting task and incorporated retention trials, quality of movement exploration, and bilateral weight shifting.

During Phase I, individuals in both groups sat unsupported on a hi-lo mat table which was adjusted so participants were sitting at 90 degrees hip and knee flexion with feet shoulder width apart. Tape marks were used to mark initial set up ensuring standardized positioning for each trial. Following baseline trials, all participants watched the same instructional video describing lateral weight shifting. The instructions included correct mechanics that should be used when weight shifting laterally with focus on correct form needed for the movement.

Testing included baseline, acquisition, short term retention (5 minutes later), and long-term retention (7-10 days later). Participants performed three trials of seated weight shifting to each side at all timepoints. During acquisition, the internal focus group was instructed to "shift your weight as much as possible towards your right or left hip without using your arms". The external focus group sat with targets one arm length away at shoulder height and were instructed to "shift your body weight as much as possible towards the blue/orange target without using your arms." During baseline and retention trials, adults were instructed to "lean as far as you can to the right/left without using your arms." During Phase II, the protocol was similar except 6 trials were performed for acquisition to potentially improve motor learning, which was not significant in Phase I per retention data. Other changes to the protocol included allowing participants to move their feet when weight-shifting. Instructions were also revised. The external focus group was told to "move your shoulder as close to the blue/orange target as possible", while the internal focus group was told to "shift your body weight as much as possible towards your right/left hip without using your arms."

ELIGIBILITY:
Inclusion Criteria:

* participants with history of stroke
* ability to sit statically without physical assistance

Exclusion Criteria:

* severe hemineglect (star cancellation test <44/54)
* inability to follow multistep commands
* orthopedic issues that limited their ability to weight shift including severe hip or back pain
* individuals with other neurologic conditions such as dementia
* individuals with contraversive pushing.

During the first arm (phase) of the study there were age matched healthy controls.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | One year for each arm of the study.
  Percentage of participants recruited out of the estimated number needed by power analysis. Power analyses revealed 42 participants were needed for 2X4 mixed model ANOVA 193 analysis, a=.05, power=.8, with a medium effect size, f=.2.
Retention | One year for each arm of the study.
  Percentage of participants that completed all 4 timepoints, baseline, acquisition, short term, and long term retention out of those that completed baseline trials.

SECONDARY OUTCOMES:
Shoulder alignment during baseline to affected side | baseline (prior to training)
  Only used in arm 2 of the study. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.
  A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during baseline to unaffected side | baseline (prior to training)
  Only used in arm 2 of the study. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.
  A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during acquisition or training to affected side | acquisition (30 minutes) through study completion, average of one year.
  Arm 2 only. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.Baseline measurements are taken, then participants are given a 2 minute demonstration of what to do during training. The training or acquisition occurs right afterwards.A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during acquisition or training to unaffected side | acquisition (30 minutes) through study completion, average of one year.
  Arm 2 only. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis. Baseline measurements are taken, then participants are given a 2 minute demonstration of what to do during training. The training or acquisition occurs right afterwards. A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during short term retention to affected side | short-term (5 minutes after training)
  Only used in arm 2 of the study. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.
  A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during short term retention to unaffected side | short-term (5 minutes after training)
  Only used in arm 2 of the study. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.
  A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during long term retention to affected side | long-term (7 days after training)
  Only used in arm 2 of the study. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.
  A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Shoulder alignment during long term retention to unaffected side | long-term (7 days after training)
  Only used in arm 2 of the study. Angle measuring a line from acromion to acromion compared to a horizontal plumb line. This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. Participants shifted to both sides 6 times to each side during arm 2 of the study. Averages were used for data analysis.
  A 9.5" X 7.31" X 0.37" 4th generation iPad†, with a 9.7-inch retina display, was used to record videos of each trial. The iPad has a 1080p HD video and 1.2 MP photo camera with autofocus and a 2.4 aperture with video stabilization. From this footage, shoulder alignment was measured during seated lateral weight shifting using the Body Align Pro app‡, trademarked on Nov. 28, 2014.
Seated lateral excursion during baseline to affected side | baseline (prior to training)
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during baseline to unaffected side | baseline (prior to training)
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during acquisition or training to affected side | acquisition (30 minutes) through study completion, average of one year.
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study. Baseline measurements are taken, then participants are given a 2 minute demonstration of what to do during training. The training or acquisition occurs right after this demonstration and occurs for 30 minutes.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during acquisition or training to unaffected side | acquisition (30 minutes) through study completion, average of one year.
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study. Baseline measurements are taken, then participants are given a 2 minute demonstration of what to do during training. The training or acquisition occurs right after this demonstration and occurs for 30 minutes.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during short-term retention to affected side | short-term (5 minutes after training)
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during short-term retention to unaffected side | short-term (5 minutes after training)
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during long-term retention to affected side | long-term (7 days after training)
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.
Seated lateral excursion during long-term retention to unaffected side | long-term (7 days after training)
  Measure of how far individuals shifted their center of pressure laterally during each weight shift trial (cm). This is a repeated measure over 4 time points. This measurement will occur during each lateral weight shift for all participants. Pt's will shift to either side 3 times during baseline, short term and long term retention. In arm 1 participants shifted to both sides 3 times during the acquisition trials and 6 times to each side during arm 2 of the study.
  A 32X32 array BodiTrak* pressure mat with an 18.125 in x 18.125 in sensing area (1,024 sensors) was used to measure lateral excursion of center of pressure during each trial for both phases. The pressure mat has a 200 mmHg calibration range and up to 150 Hz sampling frame rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley W Hyatt, DPT, Principal Investigator — Western Carolina University
Locations (1):
- Western Carolina University, Cullowhee, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Wulf G. Attentional focus and motor learning: A review of 15 years. Int Rev Sport Exerc Psychol. 2013;6(1):77-104. doi:10.1080/1750984X.2012.723728
- [Background] Kal EC, van der Kamp J, Houdijk H. External attentional focus enhances movement automatization: a comprehensive test of the constrained action hypothesis. Hum Mov Sci. 2013 Aug;32(4):527-39. doi: 10.1016/j.humov.2013.04.001. Epub 2013 Jun 30. PMID 24054892
- [Background] Kakebeeke T, Knols R, de Bruin E. Should rehabilitation specialists use external focus instructions when motor learning is fostered? A systematic review. Sports. 2013;1(2):37-54. doi:10.3390/sports1020037
- [Background] Wulf G, McNevin N, Shea CH. The automaticity of complex motor skill learning as a function of attentional focus. Q J Exp Psychol A. 2001 Nov;54(4):1143-54. doi: 10.1080/713756012. PMID 11765737
- [Background] Sturmberg C, Marquez J, Heneghan N, Snodgrass S, van Vliet P. Attentional focus of feedback and instructions in the treatment of musculoskeletal dysfunction: a systematic review. Man Ther. 2013 Dec;18(6):458-67. doi: 10.1016/j.math.2013.07.002. Epub 2013 Sep 3. PMID 24008053
- [Background] McNevin NH, Wulf G, Carlson C. Effects of attentional focus, self-control, and dyad training on motor learning: implications for physical rehabilitation. Phys Ther. 2000 Apr;80(4):373-85. doi: 10.1093/ptj/80.4.373. PMID 10758522
- [Background] Masters RSW. Knowledge, knerves and know-how: The role of explicit versus implicit knowledge in the breakdown of a complex motor skill under pressure. Br J Psychol. 1992;83:343-358.
- [Background] Kal EC, van der Kamp J, Houdijk H, Groet E, van Bennekom CA, Scherder EJ. Stay Focused! The Effects of Internal and External Focus of Attention on Movement Automaticity in Patients with Stroke. PLoS One. 2015 Aug 28;10(8):e0136917. doi: 10.1371/journal.pone.0136917. eCollection 2015. PMID 26317437
- [Background] Kal E, Houdijk H, van der Kamp J, Verhoef M, Prosee R, Groet E, Winters M, van Bennekom C, Scherder E. Are the effects of internal focus instructions different from external focus instructions given during balance training in stroke patients? A double-blind randomized controlled trial. Clin Rehabil. 2019 Feb;33(2):207-221. doi: 10.1177/0269215518795243. Epub 2018 Aug 31. PMID 30168348
- [Background] Kim GJ, Hinojosa J, Rao AK, Batavia M, O'Dell MW. Randomized Trial on the Effects of Attentional Focus on Motor Training of the Upper Extremity Using Robotics With Individuals After Chronic Stroke. Arch Phys Med Rehabil. 2017 Oct;98(10):1924-1931. doi: 10.1016/j.apmr.2017.06.005. Epub 2017 Jun 24. PMID 28652064
- [Background] Durham KF, Sackley CM, Wright CC, Wing AM, Edwards MG, van Vliet P. Attentional focus of feedback for improving performance of reach-to-grasp after stroke: a randomised crossover study. Physiotherapy. 2014 Jun;100(2):108-15. doi: 10.1016/j.physio.2013.03.004. Epub 2013 Jun 21. PMID 23796803
- [Background] Fasoli SE, Trombly CA, Tickle-Degnen L, Verfaellie MH. Effect of instructions on functional reach in persons with and without cerebrovascular accident. Am J Occup Ther. 2002 Jul-Aug;56(4):380-90. doi: 10.5014/ajot.56.4.380. PMID 12125827
- [Background] Muckel S, Mehrholz J. Immediate effects of two attention strategies on trunk control on patients after stroke. A randomized controlled pilot trial. Clin Rehabil. 2014 Jul;28(7):632-6. doi: 10.1177/0269215513513963. Epub 2014 Jan 22. PMID 24452700
- [Background] Ziv G, Lidor R. Attentional focus and motor learning in clinical settings and in older age: A review. J Mot Learn Dev. 2015;3(2):123-139. doi:10.1123/jmld.2015-0014
- [Background] Perennou DA, Mazibrada G, Chauvineau V, Greenwood R, Rothwell J, Gresty MA, Bronstein AM. Lateropulsion, pushing and verticality perception in hemisphere stroke: a causal relationship? Brain. 2008 Sep;131(Pt 9):2401-13. doi: 10.1093/brain/awn170. Epub 2008 Aug 4. PMID 18678565
- [Background] Becker K, Smith PJ. Age, task complexity, and sex as potential moderators of attentional focus effects. Percept Mot Skills. 2013 Aug;117(1):1172-86. doi: 10.2466/23.25.pms.117x14z3. PMID 24422344
- [Background] Johnson L, Burridge JH, Demain SH. Internal and external focus of attention during gait re-education: an observational study of physical therapist practice in stroke rehabilitation. Phys Ther. 2013 Jul;93(7):957-66. doi: 10.2522/ptj.20120300. Epub 2013 Apr 4. PMID 23559523
- [Background] Shafizadeh M, Platt GK, Mohammadi B. Effects of different focus of attention rehabilitative training on gait performance in Multiple Sclerosis patients. J Bodyw Mov Ther. 2013 Jan;17(1):28-34. doi: 10.1016/j.jbmt.2012.04.005. Epub 2012 May 10. PMID 23294680
- [Background] McKay B, Wulf G. A distal external focus enhances novice dart throwing performance. Int J Sport Exerc Psychol. 2012;10(2):149-156. doi:10.1080/1612197X.2012.682356
- [Background] McNevin NH, Shea CH, Wulf G. Increasing the distance of an external focus of attention enhances learning. Psychol Res. 2003 Feb;67(1):22-9. doi: 10.1007/s00426-002-0093-6. Epub 2002 Oct 30. PMID 12589447
- [Background] Kal E, van den Brink H, Houdijk H, van der Kamp J, Goossens PH, van Bennekom C, Scherder E. How physical therapists instruct patients with stroke: an observational study on attentional focus during gait rehabilitation after stroke. Disabil Rehabil. 2018 May;40(10):1154-1165. doi: 10.1080/09638288.2017.1290697. Epub 2017 Feb 24. PMID 28637152
- [Background] Lam JM, Globas C, Hosp JA, Karnath HO, Wachter T, Luft AR. Impaired implicit learning and feedback processing after stroke. Neuroscience. 2016 Feb 9;314:116-24. doi: 10.1016/j.neuroscience.2015.11.051. Epub 2015 Nov 27. PMID 26633264
- [Background] Chiviacowsky S, Wulf G, Wally R. An external focus of attention enhances balance learning in older adults. Gait Posture. 2010 Oct;32(4):572-5. doi: 10.1016/j.gaitpost.2010.08.004. Epub 2010 Sep 17. PMID 20850325
- [Background] McNevin N, Weir P, Quinn T. Effects of attentional focus and age on suprapostural task performance and postural control. Res Q Exerc Sport. 2013 Mar;84(1):96-103. doi: 10.1080/02701367.2013.762321. PMID 23611013
- See also: Founder letter : Is the 8 % payment cut the wake-up call rehab therapists need? WebPT — https://www.webpt.com/blog/post/founder-letter-is-the-8-payment-cut-the-wake-up-call-rehab-therapists-need/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04696302/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04696302/ICF_001.pdf